CLINICAL TRIAL: NCT04997954
Title: EMERALD TRIAL Open-Label Extension Study (EMERALD OLE)
Brief Title: EMERALD TRIAL Open Label Extension Study
Acronym: EMERALD-OLE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gold Coast Hospital and Health Service (Other Government)
Collaborators: Bod Australia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCMR0001-OLE
Record Dates: First submitted 2021-07-26; First posted 2021-08-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Cannabis; CBD; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Marijuana Abuse; Motor Neuron Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MediCabilis CBD Oil (Experimental): MediCabilis CBD Oil to be taken no more than 7ml/day orally based from participants' individual 14 day titration period completed at the beginning of the trial. The frequency of the drug intake can range between once and three times a day depending on the outcome of the 14 day titration period. Titration period allows participants to gradually increase study drug intake in order to find appropriate dose for participants without or with minimal undesired side effects. The treatment will last no more than 6 months.
  Interventions: Drug: MediCabilis CBD oil

INTERVENTIONS:
Drug: MediCabilis CBD oil — The investigational product (MediCabilis 5% (50mg/ml) CBD Oil) will be supplied by BOD Australia, an Australian licensed manufacturer of medical grade cannabis.
  The main components of MediCabilis 5% (50 mg/mL) CBD extract in MCT Oil are:
  * Cannabis sativa L. dry extract
  * Medium chain triglycerides (Ph Eur 0868) which are added in order to adjust the active constituent (cannabidiol) to the target content.
  Each mL of MediCabilis provides:
  * 50 mg of Cannabidiol (CBD+CBDA)
  * Less than 2 mg tetrahydrocannabinol (THC)
  * Non-active ingredient: Medium Chain Triglycerides (MCT) oil sourced from coconut

SUMMARY:
EMERALD OLE trial is an open-label extension of the EMERALD trial. Long term tolerability and safety of the MediCabilis CBD oil has not been extensively studied. EMERALD OLE aims to establish data on the prolonged used of the study drug product.

All participants who completed the EMERALD trial will be offered to enter EMERALD OLE. Participants will be taking the active drug MediCabilis CBD oil for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS/MND, either definite or probable according to the El Escorial revised criteria
* Can provide written informed consent
* Able and willing to comply with all study requirement
* Male or female, 25-80 years old
* Randomised into the EMERALD trial

Exclusion Criteria:

* Participants who are bedridden
* History of any psychiatric disorder other than depression associated with their underlying condition including immediate family history of schizophrenia
* Heavy consumption of alcohol or use of illicit drug
* Hypersensitivity to cannabinoids or any of the excipients
* Any of the following: eGFR <30 mL/min/1.73m2, ejection fraction <35%, or AST and ALT >5 X ULN
* Unwillingness of a female participant of child-bearing potential, or their partner, to use effective contraception during the study and 30 days thereafter
* Pregnant, lactating mother or female participant planning pregnancy during the course of the study and for 30 days thereafter
* Received any investigational drug or medical device within 30 days prior randomisation except MediCabilis CBD Oil
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study
* Inability to cooperate with the study procedures
* Unwilling to stop driving vehicle or operating dangerous machinery whilst on study drug.
* Close affiliation with the study team, e.g. close relative of the investigator

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events [safety and tolerability]. | 6 months
  AE collection

SECONDARY OUTCOMES:
To evaluate the long-term effects of MediCabilis CBD Oil on the functional status of MND patients using Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) | 6 months
  Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS-R) scale will be used to assess this outcome. Minimum score: 0, Maximum score: 48. Higher scores mean better outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Gold Coast Hospital and Health Service, Gold Coast, Queensland, Australia